CLINICAL TRIAL: NCT02473055
Title: A Randomized Controlled Trial of Kangaroo Care (Skin-to-Skin) Effects on Sleep in Premature Infants
Brief Title: Kangaroo Care and Premature Infant Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Susan Ludington, Walters Professor of Pediatric Nursing, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KangarooCareEEG
Record Dates: First submitted 2015-06-10; First posted 2015-06-16 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Premature Birth of Newborn
Keywords: kangaroo care; sleep; heart rate; respiratory rate; preterm infant
MeSH Terms: conditions — Premature Birth | interventions — Kangaroo-Mother Care Method

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Kangaroo care (Experimental): kangaroo Care was skin-to-skin, chest-to-chest placement of preterm infant wearing only a diaper placed up against mother's chest and covered in one receiving blanket folded into fourth
  Interventions: Other: Kangaroo Care
- control (No Intervention): control infants remained prone in an incubator wearing only diaper

INTERVENTIONS:
Other: Kangaroo Care — skin-to-skin, chest-to-chest placement of diaper clad preterm infant up against his mother's chest and covered by a receiving blanket folded into fourths for 2-3 hours from one feeding to the next.
  Other Names: skin-to-skin contact
  Arms: Kangaroo care

SUMMARY:
90 preterm infants were randomly assigned to kangaroo care (skin-to-=skin, chest-to-chest) group (n=50) or control (remained in incubator, prone (n=40) for a pretest period of 2- 3 hours, then fed, then KC group was placed in KC and control group remained in incubator for a 2-3 hr test period. EEG measures of sleep, HR, and RR were taken. .

DETAILED DESCRIPTION:
The neonatal intensive care unit (NICU) environment is not conducive to sleep, and infant sleep in incubators is fragmented. Sleep contributes to brain maturation so interventions to foster sleep are needed. During Kangaroo Care (KC) behavioral indicators of Quiet Sleep have been observed but, not confirmed by objective electroencephalographic (EEG) analysis.The purpose was to determine the effects of Kangaroo Care (KC) on EEG-based sleep using Nihon Koden polysomnography and cardiorespiratory patterns by comparing KC sleep to incubator sleep.. A randomized controlled study with 90 preterms (KC = 50; control = 40) in which KC infants received 2-3 hours of KC between feeds after a comparable pretest period in an incubator and control infants remained in an incubator during the 2-3 hour pretest and test periods. In the incubator infants were inclined, prone, and nested; in KC infants were inclined, prone, and chest-to-chest underneath a blanket. The medically stable preterm infants were a mean 32 weeks postmenstrual age.

ELIGIBILITY:
Inclusion Criteria:

* Subjects whose five-minute APGARS were greater than 6, gestational age was 28 or more weeks at birth, and whose testing weight was greater than 1000 grams were included.

Exclusion Criteria:

* Infants with encephalopathy, intraventricular hemorrhage greater than grade II, white matter lucencies on cranial ultrasound, seizures, meningitis, or congenital brain malformations were excluded

Ages: 7 Days to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2003-01; Primary Completion 2008-06 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
EEG-based sleep | 2-3 hours
  Infants attached to EEG machine and Respiratory impedance plethysmography bands prior to beginning of pretest period and remainded on EEG until end of study

SECONDARY OUTCOMES:
Heart rates during pretest | 2-3 hours of pretest
  Heart Rate was detected by Nihon Koden polysomnograph
Respiratory rate during pretest | 2-3 hours pretest
  Impedance plethysmography belts attached to Nihon Koden polysomnograph machine
Heart rates during test | 2-3 hours of test
  Heart rate was detected by Nihon Koden polysomnograph
Respiratory rate during test period | 2-3 hours test period
  Impedance plethysmography belts attached to Nihon Koden polysomnograph machine

CONTACTS AND LOCATIONS:
Overall Officials: Susan Ludington, Principal Investigator — Case Western Reserve University Frances Payne Bolton School of Nursing
Locations (1):
- UH hospitals, Cleveland, Ohio, United States

REFERENCES:
- [Background] Mazurier E, Picaud JC. [Kangaroo mother care vs nidcap: a problem of semantics]. Arch Pediatr. 2005 Apr;12(4):471-2; author reply 473. doi: 10.1016/j.arcped.2004.12.019. No abstract available. French. PMID 15808441
- [Background] Als H, Duffy FH, McAnulty GB, Rivkin MJ, Vajapeyam S, Mulkern RV, Warfield SK, Huppi PS, Butler SC, Conneman N, Fischer C, Eichenwald EC. Early experience alters brain function and structure. Pediatrics. 2004 Apr;113(4):846-57. doi: 10.1542/peds.113.4.846. PMID 15060237
- [Background] Perlman JM. The genesis of cognitive and behavioral deficits in premature graduates of intensive care. Minerva Pediatr. 2003 Apr;55(2):89-101. PMID 12754453
- [Background] Whitney MP, Thoman EB. Early sleep patterns of premature infants are differentially related to later developmental disabilities. J Dev Behav Pediatr. 1993 Apr;14(2):71-80. PMID 7682580
- [Background] Holditch-Davis D, Scher M, Schwartz T, Hudson-Barr D. Sleeping and waking state development in preterm infants. Early Hum Dev. 2004 Oct;80(1):43-64. doi: 10.1016/j.earlhumdev.2004.05.006. PMID 15363838
- [Background] Scher MS, Sun M, Steppe DA, Banks DL, Guthrie RD, Sclabassi RJ. Comparisons of EEG sleep state-specific spectral values between healthy full-term and preterm infants at comparable postconceptional ages. Sleep. 1994 Feb;17(1):47-51. doi: 10.1093/sleep/17.1.47. PMID 8191202
- [Background] Sesma HW, Georgieff MK. The effect of adverse intrauterine and newborn environments on cognitive development: the experiences of premature delivery and diabetes during pregnancy. Dev Psychopathol. 2003 Fall;15(4):991-1015. doi: 10.1017/s0954579403000488. PMID 14984135
- [Background] Pillai M, James D. Behavioural states in normal mature human fetuses. Arch Dis Child. 1990 Jan;65(1 Spec No):39-43. doi: 10.1136/adc.65.1_spec_no.39. PMID 2306133
- [Background] Mirmiran M, Maas YG, Ariagno RL. Development of fetal and neonatal sleep and circadian rhythms. Sleep Med Rev. 2003 Aug;7(4):321-34. doi: 10.1053/smrv.2002.0243. PMID 14505599
- [Background] Feldman R, Eidelman AI. Skin-to-skin contact (Kangaroo Care) accelerates autonomic and neurobehavioural maturation in preterm infants. Dev Med Child Neurol. 2003 Apr;45(4):274-81. doi: 10.1017/s0012162203000525. PMID 12647930
- [Background] Mestyan J, Jarai I, Fekete M. The total energy expdenditure and its components in premature infants maintained under different nursing and environmental conditions. Pediatr Res. 1968 May;2(3):161-71. doi: 10.1203/00006450-196805000-00002. No abstract available. PMID 5659088
- [Background] Spangler G, Scheubeck R. Behavioral organization in newborns and its relation to adrenocortical and cardiac activity. Child Dev. 1993 Apr;64(2):622-33. PMID 8477638
- [Background] Peirano P, Algarin C, Uauy R. Sleep-wake states and their regulatory mechanisms throughout early human development. J Pediatr. 2003 Oct;143(4 Suppl):S70-9. doi: 10.1067/s0022-3476(03)00404-9. PMID 14597916
- [Background] Ohgi S, Arisawa K, Takahashi T, Kusumoto T, Goto Y, Akiyama T, Saito H. Neonatal behavioral assessment scale as a predictor of later developmental disabilities of low birth-weight and/or premature infants. Brain Dev. 2003 Aug;25(5):313-21. doi: 10.1016/s0387-7604(02)00233-4. PMID 12850509
- [Background] Vertes RP, Eastman KE. The case against memory consolidation in REM sleep. Behav Brain Sci. 2000 Dec;23(6):867-76; discussion 904-1121. doi: 10.1017/s0140525x00004003. PMID 11515146
- [Background] OURTH L, BROWN KB. Inadequate mothering and disturbance in the neonatal period. Child Dev. 1961 Jun;32:287-95. doi: 10.1111/j.1467-8624.1961.tb05026.x. No abstract available. PMID 13731731
- [Background] Ludington-Hoe SM, Anderson GC, Swinth JY, Thompson C, Hadeed AJ. Randomized controlled trial of kangaroo care: cardiorespiratory and thermal effects on healthy preterm infants. Neonatal Netw. 2004 May-Jun;23(3):39-48. doi: 10.1891/0730-0832.23.3.39. PMID 15182119
- [Background] Brazy JE, Goldstein RF, Oehler JM, Gustafson KE, Thompson RJ Jr. Nursery neurobiologic risk score: levels of risk and relationships with nonmedical factors. J Dev Behav Pediatr. 1993 Dec;14(6):375-80. PMID 8126229
- [Background] Ludington-Hoe SM, Johnson MW, Morgan K, Lewis T, Gutman J, Wilson PD, Scher MS. Neurophysiologic assessment of neonatal sleep organization: preliminary results of a randomized, controlled trial of skin contact with preterm infants. Pediatrics. 2006 May;117(5):e909-23. doi: 10.1542/peds.2004-1422. PMID 16651294
- [Background] Scher MS, Jones BL, Steppe DA, Cork DL, Seltman HJ, Banks DL. Functional brain maturation in neonates as measured by EEG-sleep analyses. Clin Neurophysiol. 2003 May;114(5):875-82. doi: 10.1016/s1388-2457(03)00026-9. PMID 12738433
- [Background] Lehtonen L, Martin RJ. Ontogeny of sleep and awake states in relation to breathing in preterm infants. Semin Neonatol. 2004 Jun;9(3):229-38. doi: 10.1016/j.siny.2003.09.002. PMID 15050216
- [Background] Gerard CM, Harris KA, Thach BT. Spontaneous arousals in supine infants while swaddled and unswaddled during rapid eye movement and quiet sleep. Pediatrics. 2002 Dec;110(6):e70. doi: 10.1542/peds.110.6.e70. PMID 12456937
- [Background] Franco P, Scaillet S, Valente F, Chabanski S, Groswasser J, Kahn A. Ambient temperature is associated with changes in infants' arousability from sleep. Sleep. 2001 May 1;24(3):325-9. doi: 10.1093/sleep/24.3.325. PMID 11322716
- [Background] Horne RS, Bandopadhayay P, Vitkovic J, Cranage SM, Adamson TM. Effects of age and sleeping position on arousal from sleep in preterm infants. Sleep. 2002 Nov 1;25(7):746-50. doi: 10.1093/sleep/25.7.746. PMID 12405610
- [Background] White-Traut RC, Pate CM. Modulating infant state in premature infants. J Pediatr Nurs. 1987 Apr;2(2):96-101. No abstract available. PMID 3550039
- [Background] Lacy JB, Ohlsson A. Behavioral outcomes of environmental or care-giving hospital-based interventions for preterm infants: a critical overview. Acta Paediatr. 1993 Apr;82(4):408-15. doi: 10.1111/j.1651-2227.1993.tb12709.x. No abstract available. PMID 8318812
- [Background] Fransson AL, Karlsson H, Nilsson K. Temperature variation in newborn babies: importance of physical contact with the mother. Arch Dis Child Fetal Neonatal Ed. 2005 Nov;90(6):F500-4. doi: 10.1136/adc.2004.066589. PMID 16244210
- [Background] Schrod L, Walter J. Effect of head-up body tilt position on autonomic function and cerebral oxygenation in preterm infants. Biol Neonate. 2002;81(4):255-9. doi: 10.1159/000056756. PMID 12011569
- [Background] Tuladhar R, Harding R, Michael Adamson T, Horne RS. Comparison of postnatal development of heart rate responses to trigeminal stimulation in sleeping preterm and term infants. J Sleep Res. 2005 Mar;14(1):29-36. doi: 10.1111/j.1365-2869.2004.00434.x. PMID 15743331
- [Background] Tornhage CJ, Stuge E, Lindberg T, Serenius F. First week kangaroo care in sick very preterm infants. Acta Paediatr. 1999 Dec;88(12):1402-4. doi: 10.1080/080352599750030167. PMID 10626530
- [Background] Franco P, Seret N, Van Hees JN, Lanquart JP Jr, Groswasser J, Kahn A. Cardiac changes during sleep in sleep-deprived infants. Sleep. 2003 Nov 1;26(7):845-8. doi: 10.1093/sleep/26.7.845. PMID 14655918